CLINICAL TRIAL: NCT04967781
Title: Autoimmunity Contributes to the Severe Progression of COVID-19
Status: Completed | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AUTO001
Record Dates: First submitted 2021-07-13; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Coronavirus Disease 2019
MeSH Terms: conditions — COVID-19 | interventions — Autoimmunity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group "Severe": Each enrolled patient was allocated into control group "Non-severe" or case group "Severe" as per the disease severity which was defined according to the Chinese novel coronavirus pneumonia prevention and control guideline (version 6.0), "severe" and "critical" types were grouped into case group as "Severe".
  Interventions: Behavioral: autoimmunity
- Group "Non-severe": Each enrolled patient was allocated into control group "Non-severe" or case group "Severe" as per the disease severity which was defined according to the Chinese novel coronavirus pneumonia prevention and control guideline (version 6.0), "mild" and "moderate" types were grouped into control group as "Non-severe".

INTERVENTIONS:
Behavioral: autoimmunity — autoimmunity is characterized as self attacking from self immune system, which may involve in the severe progression of COVID-19.
  Groups: Group "Severe"

SUMMARY:
Although elderliness and chronic comorbidities such as hypertension, diabetes, cardiovascular diseases and respiratory diseases, are known risk factors for severe progression of COVID-19, it still remains puzzling on why younger patients without any comorbidity advance to severity and even more rapidly, the underlying mechanisms for severe progression of COVID-19 still needs to be elucidated. Based on current picturing of the COVID-19, similar to SARS, besides direct viral toxicity, immune-mediated attack derived from either the release of pro-inflammatory cytokine perpetual cascade, or secondary pathogen-induced autoimmunity response may also play important roles on disease progression and partly account for the multi-system injuries related with COVID-19. Virus infection has been implicated in the initiation of autoimmunity, which can attack multiple systems. With the knowledge of characteristics of SARS, high level of autoimmune activity was shown to make severe injuries to lungs or other organs, leading to poor outcome including multi-system failure9. COVID-19 may also get autoimmunity involved which is of obviously younger and female population predominance during the pathogenesis, no matter pre-existing or secondary to viral infection. Particularly strong immune response to SARS-CoV-2 infection might not be protective, but perhaps, be harmful to the host, contributing to disease severe progression.

ELIGIBILITY:
Inclusion Criteria:

1. Adult inpatients from two centers, Zhongnan Hospital of Wuhan University and Thunder God Mountain Hospital, Wuhan, China.
2. Experimental confirmed COVID-19 patients.
3. Patients tested with autoimmunological detections including either ANA+ENA (Antinuclear antibody + Anti-extractable nuclear antigen antibody), Anti-cardiolipin antibody (ACA), Rheumatoid factor (RF), or Anti-streptolysin O antibody (ASO) detection.

Exclusion Criteria:

1. Minors.
2. Experimental un-confirmed COVID-19 patients.
3. Patients without autoimmunological detections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The retrospective study includes two groups of adult inpatients from two centers, Zhongnan Hospital of Wuhan University and Thunder God Mountain Hospital, Wuhan, China. All patients who were diagnosed as COVID-19 with real-time PCR (RT-PCR) assay of pharyngeal swab specimens18 confirmed results were screened, and those tested with autoimmunological detections including either ANA+ENA (Antinuclear antibody + Anti-extractable nuclear antigen antibody), Anti-cardiolipin antibody (ACA), Rheumatoid factor (RF), or Anti-streptolysin O antibody (ASO) detection, were enrolled in our study from Jan 22, 2020 to Jun 24, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Presence of Antinuclear autoantibodies detected by ANA+ENA test | baseline
  Antinuclear antibodies are closely related with many autoimmune diseases, and involved in the pathogenesis of many kinds of viruses.ANA+ENA was subjected to test from the admission till the discharge of patients' hospitalization. Both positive and negative results were reported, and detailed specific autoantibodies were also reported if positive.
Presence of Antinuclear autoantibodies detected by ANA+ENA test | from the admission till the discharge of patients' hospitalization, up to 100 days.
  Antinuclear antibodies are closely related with many autoimmune diseases, and involved in the pathogenesis of many kinds of viruses.ANA+ENA was subjected to test from the admission till the discharge of patients' hospitalization. Both positive and negative results were reported, and detailed specific autoantibodies were also reported if positive.
Presence of Anti-streptolysin O (ASO) | baseline
  Anti-streptolysin O (ASO or ASLO) is the antibody made against streptolysin O, an immunogenic, oxygen-labile hemolytic toxin produced by most strains of group A and many strains of groups C and G streptococci.ASO was subjected to test from the admission till the discharge of patients' hospitalization. Both positive and negative results were reported, and detailed specific immune globulin types were also reported if positive.
Presence of Anti-streptolysin O (ASO) | from the admission till the discharge of patients' hospitalization, up to 100 days.
  Anti-streptolysin O (ASO or ASLO) is the antibody made against streptolysin O, an immunogenic, oxygen-labile hemolytic toxin produced by most strains of group A and many strains of groups C and G streptococci.ASO was subjected to test from the admission till the discharge of patients' hospitalization. Both positive and negative results were reported, and detailed specific immune globulin types were also reported if positive.
Presence of Rheumatoid Factors (RF) | baseline
  factors used for the diagnosis of the rheumatoid arthritis (RA).RF was subjected to test from the admission till the discharge of patients' hospitalization. Both positive and negative results were reported, and detailed specific immune globulin types were also reported if positive.
Presence of Rheumatoid Factors (RF) | From the admission till the discharge of patients' hospitalization, up to 100 days.
  factors used for the diagnosis of the rheumatoid arthritis (RA).RF was subjected to test from the admission till the discharge of patients' hospitalization. Both positive and negative results were reported, and detailed specific immune globulin types were also reported if positive.
Presence of Anticardiolipin antibody (ACA) | baseline
  Anti- cardiolipin antibody (ACA) targets against anionic phospholipids and inhibits the effect of the prothrombin-activator complex to cause arterial and/or venous thrombosis, transiently appears positive around times of acute infections and acute thrombosis.ACA was subjected to test from the admission till the discharge of patients' hospitalization. Both positive and negative results were reported, and detailed specific immune globulin types were also reported if positive.
Presence of Anticardiolipin antibody (ACA) | From the admission till the discharge of patients' hospitalization, up to 100 days.
  Anti- cardiolipin antibody (ACA) targets against anionic phospholipids and inhibits the effect of the prothrombin-activator complex to cause arterial and/or venous thrombosis, transiently appears positive around times of acute infections and acute thrombosis.ACA was subjected to test from the admission till the discharge of patients' hospitalization. Both positive and negative results were reported, and detailed specific immune globulin types were also reported if positive.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
With the permission of the corresponding author, we can provide participant data without names and identifiers, but not the study protocol, statistical analysis plan, or informed consent form. Data can be provided after the article is published. Once the data can be made public, the research team will provide an email address for communication. The corresponding authors have the right to decide whether to share the data or not based on the research objectives and plan provided.